CLINICAL TRIAL: NCT01858350
Title: Comparison of the Effectiveness of Complementary and Alternative Medicine (CAM) Therapies in Pediatric Patients Undergoing Medical Resonance Imagining (MRI) Studies
Brief Title: Comparison of the Effectiveness of CAM Therapies in Pediatric Patients Undergoing Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Ambika Mathur, Professor, Wayne State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC1AT005699 (NIH)
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Neurological Disorders
Keywords: CAM; Sedation; MRI; Music Therapy
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active Music Therapy (Other): Active Music Therapy: A music therapist plays music to patients for 15 minutes
  Interventions: Other: Active Music Therapy
- Passive Music Therapy (Other): Passive Music Therapy: A music therapist plays a compact disc (CD) to patients for 15 minutes
  Interventions: Other: Passive Music Therapy
- No intervention (No Intervention)
- Distraction Therapy (Other): Distraction Therapy: A child life specialist plays with patients for 15 minutes
  Interventions: Other: Distraction Therapy

INTERVENTIONS:
Other: Active Music Therapy
  Arms: Active Music Therapy
Other: Passive Music Therapy
  Arms: Passive Music Therapy
Other: Distraction Therapy
  Arms: Distraction Therapy

SUMMARY:
The investigators conducted a prospective open unblinded clinical four-arm evaluation of Complementary and Alternate Medicine (CAM) interventions on children 1-12 years of age who were undergoing imaging by Medical Resonance Imaging(MRI) and receiving parenteral sedation. Children were assigned to active music therapy, passive music therapy, distraction therapy, and no intervention; measures included doses and numbers of sedation medications, time of sedation, and salivary levels of the stress hormone cortisol and pro-inflammatory cytokines, before and immediately after the intervention was completed. The Time Frame for the outcome measures are at the start of the intervention and immediately following the procedure (generally about 150 minutes). No further follow up was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 1-12 years undergoing MRI studies

Exclusion Criteria:

* Patients with significant congenital anomalies, genetic syndromes and central nervous system malformations

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 471 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Need for sedation medications for MRI is reduced | The Time Frame for the outcome measures are at the start of the intervention and immediately following the procedure (average about 150 minutes). No further follow up was conducted.
  Intervention is performed prior to sedation. Following sedation, the patient undergoes MRI. After the MRI is completed, the amount of sedation given to the patient is recorded. No other follow up is required.

SECONDARY OUTCOMES:
To measure the effect of the interventions on salivary cortisol and inflammatory cytokines | Saliva samples were collected before the intervention and then after the MRI was performed (average about 150 minutes).
  The aim of this measure was to determine if the interventions changed the levels of salivary cortisol and inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Ambika MATHUR, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University and Children's Hospital of Michigan, Detroit, Michigan, United States